CLINICAL TRIAL: NCT05679622
Title: Repeated and Multiple Fecal Microbiota Transplantations in Active Pediatric Ulcerative Colitis (UC)
Brief Title: Fecal Microbiota Transplantation in Pediatric Ulcerative Colitis (UC)
Acronym: FMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biao Zou (Other)
Responsible Party: Sponsor-Investigator, Biao Zou, attending physician, Pediatric Department, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63639979
Record Dates: First submitted 2022-12-25; First posted 2023-01-11 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Ulcerative Colitis
Keywords: Fecal microbiota transplantation, Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT group (Experimental): In the refractory ulcerative colitis group, our study is aims to explore repeated and multiple FMTs plus PEN in the treatment of refractory pediatric UC;
  Interventions: Other: Fecal Microbiota Transplantation

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — In the induction stage of UC, FMT group received FMT and PEN intervention, and FMT group are given for at least one course of FMT treatment. If repeated FMTs are received, it is usually at a 2 month interval. All the participants received PEN (80% of total calories as a polymeric diet, Peptamen, Nestle, Vevey, and Switzerland) intervention to help induce and maintain clinical remission.

SUMMARY:
This study included two topics: one was to test the efficacy and safety of fecal microbiota transplants plus partial enteral nutrition (PEN) in refractory pediatric UC where conventional therapy has failed, and the other was to explore the efficacy and safety of FMT plus PEN as first-line therapy for pediatric active UC

DETAILED DESCRIPTION:
Recent studies have suggested that gut imbalance and deregulation of immunological responses plays a pivotal role in the disease development of UC, and that FMT could be a useful treatment. In the refractory ulcerative colitis group, our study is aims to explore FMT plus PEN in the treatment of refractory pediatric UC. In the induction stage of UC, standard therapy remained unchanged, FMT and PEN treatment are added, and the investigators hope the withdrawal of conventional drug therapy was gradually reduced. Refractory UC is defined as refractory to standard therapy (e.g., steroids, immunomodulators, cyclosporine, tacrolimus, or anti-TNF agents).

As a first-line treatment group for UC, our study is aims to explore FMT plus PEN as a first-line treatment for active UC in children. participants treated with FMT coupled with PEN are defined as the FMT group, and those treated with PEN coupled with mesalazine served as the PEN group.

FMT treatment is given for at least one course of FMT treatment. If repeated FMTs are received, it is usually at a 2 month interval.

All the participants received PEN (80% of total calories as a polymeric diet, Peptamen, Nestle, Vevey, and Switzerland) intervention to help induce and maintain clinical remission.

ELIGIBILITY:
Inclusion Criteria:

age of older than 2 years and younger than 16 years with no genetic diseases; as a first-line treatment group for UC, newly diagnosed with mild-to-moderate UC (defined by the PUCAI of >10 and≤64); In the refractory ulcerative colitis group, all refractory pediatric with mild-to-moderate UC (defined by the PUCAI of >10 and≤64) defined by children who failed conventional treatment (hormone, immunosuppressant, biologics); agree to received regularly colonoscopy

Exclusion Criteria:

Children who were treated by PEN (80%) less than 8 weeks; As a first-line treatment group for UC, patients who were treated with corticosteroids, methotrexate, thiopurines, and anti-TNF agents as their first-line treatment; Known contraindication to all FMT infusion method such as nasoduodenal tube insertion, oesophago-gastro-duodenoscopy (OGD), enteroscopy, colonoscopy, enema and Fecal capsule; Unwilling to give informed consent/ assent

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
clinical response | 8-12 weeks after FMT
  reduction in the Pediatric Ulcerative Colitis Activity Index (PUCAI) ≥30% from baseline
clinical remission | 8-12 weeks after FMT
  Clinical remission defined as a PUCAI <10
safety of FMT | 8-12 weeks after FMT
  All possible adverse events: fever, abdominal pain, infectious diseases and others.

SECONDARY OUTCOMES:
Number of patients requiring escalation of medical therapies | 8-12 weeks after FMT
  Number of patients requiring escalation of medical therapies based on clinical relapse. Clinical relapse is defined by requiring additional medical therapy.
Number of patients with endoscopic remission | 8-12 weeks after FMT
  Number of patients with endoscopic remission as defined by a PUCAI score of 0
Fecal calprotectin level | 8-12 weeks after FMT
  Mean change of Fecal calprotectin levels
C-reactive protein levels | 8-12 weeks after FMT
  Mean change of C-reactive protein levels
erythrocyte sedimentation rate (ESR) level | 8-12 weeks after FMT
  Mean change of erythrocyte sedimentation rate (ESR)
The number of stools or bloody stools | 8-12 weeks after FMT
  Improvement in the number of stools or bloody stools
gut microbial | before treatment and 4 weeks after treatment
  Fecal 16S RNA or macrogene sequencing was performed. Fecal samples were obtained from donor and recipient. The fecal samples and isolated microbiota samples were frozen immediately and underwent DNA extraction using standard methods.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Huang, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No